CLINICAL TRIAL: NCT01928355
Title: Cognitive Dysfunction in People Who Are Obese But Metabolically Healthy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Assy Nimer, Proffessor, Ziv Hospital
Other Study IDs: 0051-13-ziv
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- metabolically healthy
- Unhealthy

SUMMARY:
There is some evidence to suggest that obesity is a risk factor for the development of cognitive dysfunction, although this is not a universal finding. This discordance might be ascribed to the existence of a 'healthy obese phenotype'- that is, obesity in the absence of metabolic risk factors. We examined whether the association of obesity with cognitive dysfunction is dependent on the individual's metabolic health.

60 obese patients' undergoping liver fibroscan and blood tests will be enrolled. Obesity was defined as body mass index ≥ 30 kg/m2. Based on blood pressure, HDL-cholesterol, triglycerides, glycated haemoglobin, and C-reactive protein, participants were classified as 'metabolically healthy' (0 or 1 metabolic abnormality) or 'unhealthy' (≥ 2 metabolic abnormalities). Cognitive dysfunction will be assessed by moca and minimental score. Results: Cognitive dysfunction prevalence is expected in 30% , but 50% of this group was categorized as metabolically healthy. Relative to non-obese healthy participants, after adjustment for baseline covariates, the metabolically unhealthy obese participants had elevated risk of cognitive dysfunction although the metabolically healthy obese did not. The association between obesity and risk of cognitive dysfunction appears to be partly dependent on metabolic health, although further work is required to confirm these findings.

In obesity there is an increase in oxidative stress due to metabolic syndrome . Thus obese patients suffer from higher incidences of cardiovascular complications such as atherosclerosis as compare to non- obese population. Haptoglobin (Hp) is a plasma protein which binds free hemoglobin and prevents it from heme- iron mediated oxidation. There are three different types of Hp which differ in their antioxidant ability. Several clinical studies have shown that Hp 2-2 genotype is associated with higher incidence of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

Freely given written informed consent BMI>=30

Exclusion Criteria:

Evidence of Chronic Liver Diseases Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with greater body mass index
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Transient elastography | Baseline